CLINICAL TRIAL: NCT03943745
Title: Assessment of EEG Changes During Induction of Propofol Anesthesia Using Wireless Measurement Devices
Brief Title: EEG Changes During Induction of Propofol Anesthesia
Acronym: PropoStatus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: South Carelia Central Hospital (Other); Cerenion Oy (Industry)
Responsible Party: Sponsor
Other Study IDs: 31/2018
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Anesthesia, General; Healthy Subjects
Keywords: EEG; Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PropoStatus is a prospective observational study investigating the EEG changes seen in neurologically healthy patients during induction of general anesthesia with propofol.

DETAILED DESCRIPTION:
PropoStatus is a prospective observational study investigating the EEG changes seen in neurologically healthy patients during induction of general anesthesia with propofol. EEG changes are investigated in different levels of anesthesia from awake state to deep anesthesia in which burst suppression pattern (BSP) is seen in the EEG. Furthermore, the relation of EEG changes and clinically evaluated depth of anesthesia is studied.

The study population is comprised of neurologically healthy individuals who come to the hospital for elective surgery requiring general anesthesia. The patients will not receive any pre-medication. They will give a written consent to participate to the study. During induction of anesthesia, the vital signs will be monitored using the standard protocol of the operating room. EEG will be recorded using a wireless measurement device. The EEG is observed during the recording from a laptop or tablet computer. The anesthesia is induced using propofol with a fixed infusion rate of 30 mg/kg/h. The patient is asked to squeeze the anesthetist's hand repeatedly every 10 s. The moment at which the patients does not respond to the command anymore is considered as the loss of consciousness. The infusion is continued until BSP is observed in the EEG. The infusion is then continued for 3 min after which the recording of EEG is stopped. The administration of anesthesia is then continued as required by the operation.

The EEG recording will be carried out using two different devices. The first dataset, including 20 patients, will be collected using Bittium BrainStatus EEG electrode and device. The second dataset, including 30 patients, will be collected using Nihon Kohden CerebAir device.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 (no neurological or cardiovascular diseases)

Exclusion Criteria

* BMI > 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurologically healthy individuals coming to hospital for elective surgery with general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
EEG slow-wave activity | Induction of anesthesia (approx. 10-30 min)
  EEG slow-wave activity is defined by the low-frequency (<1 Hz) signal power. The study investigates the topographic distribution of the activity as well as the coupling of the activity between the electrodes. The relation of slow-wave activity and loss of consciousness will be investigated as well.

SECONDARY OUTCOMES:
EEG activity on other frequency bands | Induction of anesthesia (approx. 10-30 min)
  In addition to slow wave activity, the study investigates the topographic distribution of the activities on other frequency bands (delta, theta, alpha, beta) as well as the coupling of these activities between the electrodes.The relation of these other activities and loss of consciousness will be investigated as well.

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Kortelainen, MD, PhD, Principal Investigator — University of Oulu
Locations (1):
- South Karelia Central Hospital, Lappeenranta, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kortelainen J, Vayrynen E, Huuskonen U, Laurila J, Koskenkari J, Backman JT, Alahuhta S, Seppanen T, Ala-Kokko T. Pilot Study of Propofol-induced Slow Waves as a Pharmacologic Test for Brain Dysfunction after Brain Injury. Anesthesiology. 2017 Jan;126(1):94-103. doi: 10.1097/ALN.0000000000001385. PMID 27749312
- [Background] Kortelainen J, Vayrynen E, Juuso I, Laurila J, Koskenkari J, Ala-Kokko T. Forehead electrodes sufficiently detect propofol-induced slow waves for the assessment of brain function after cardiac arrest. J Clin Monit Comput. 2020 Feb;34(1):105-110. doi: 10.1007/s10877-019-00282-3. Epub 2019 Feb 20. PMID 30788811
- [Background] Kortelainen J, Ala-Kokko T, Tiainen M, Strbian D, Rantanen K, Laurila J, Koskenkari J, Kallio M, Toppila J, Vayrynen E, Skrifvars MB, Hastbacka J. Early recovery of frontal EEG slow wave activity during propofol sedation predicts outcome after cardiac arrest. Resuscitation. 2021 Aug;165:170-176. doi: 10.1016/j.resuscitation.2021.05.032. Epub 2021 Jun 7. PMID 34111496